CLINICAL TRIAL: NCT01022879
Title: Pain Scale in the Use of Topical Anesthesia in Small Gauge Vitrectomy
Brief Title: Topical Anesthesia in Small Gauge Vitrectomy
Acronym: Anesthesia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: APEC0004
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Pain scale of pain
MeSH Terms: conditions — Pain | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: vitrectomy

SUMMARY:
The use of topical anesthetics is a non invasive option avoiding local or general anesthesia in small gauge vitrectomy without causing intolerable pain

ELIGIBILITY:
Inclusion Criteria:

* Pseudofaquic or faquic,
* male or female,
* 18 to 80 years,
* primary vitrectomy

Exclusion Criteria:

* Combined surgery
* Non cooperative patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Martinez-Castellanos, MD, Principal Investigator — Asociación para Evitar la Ceguera en México